CLINICAL TRIAL: NCT06078007
Title: Effectiveness of a Guided Mobile App Intervention for Depression and Anxiety in University Students: a Multicenter Randomized Controlled Trial (PROMES-U Study)
Brief Title: Effectiveness of a Guided Mobile App Intervention for Depression and Anxiety in University Students (PROMES-U Study)
Acronym: PROMES-U
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Collaborators: Hospital del Mar Research Institute (IMIM) (Other); Universitat Jaume I (Other); Universidad Miguel Hernandez de Elche (Other); Universitat Pompeu Fabra (Other); Universidad de Zaragoza (Other); University of Malaga (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI20/00006; 2020/9198/I (Other: INSTITUTO DE SALUD CARLOS III)
Record Dates: First submitted 2023-09-28; First posted 2023-10-11 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Depressive Symptoms; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MyMoodCoach Intervention (Experimental)
  Interventions: Behavioral: MyMoodCoach
- Treatment-as-usual monitoring control group (No Intervention)

INTERVENTIONS:
Behavioral: MyMoodCoach — The MyMoodCoach prevention intervention is an evidence-based online intervention based on cognitive-behavioral therapy principles such as behavioral activation, problem solving and challenging negative thoughts.
  Arms: MyMoodCoach Intervention

SUMMARY:
Background: Symptoms of depression and anxiety are prevalent among Spanish university students. Minimally guided online interventions have shown promise in reducing symptomatology and preventing increased mental distress. There is a need to evaluate the effectiveness of guided preventive mental health interventions for depression and anxiety in university students.

Methods: two-arm multicenter randomized controlled trial (RCT), addressed to undergraduate students from 6 public universities with symptoms of depression and/or anxiety. Students will be evaluated through an online survey assessing mental health problems, use of mental health services, sociodemographic variables, self-perceived health, childhood and adolescent adversities, recent stressful events, social networks, personality and university experiences. A total of 600 students will be randomly assigned to: intervention group (guided E-health prevention intervention) or control group (treatment as usual with self-monitoring). The intervention, in app format, is based on principles of cognitive behavioral therapy, includes weekly feedback based on content and participation from a psychologist and self-monitoring. Assessments will take place post-intervention (up to 6 weeks), at 6 months and 12 months after randomization. The primary outcome will be the reduction of depressive or anxiety symptoms post-intervention, assessed with the Patient Health Questionnaire-9 (PHQ-9), the Generalized Anxiety Disorder-7 (GAD-7) and the Patient Health Questionnaire-Anxiety and Depression Scale (PHQ-ADS). Secondary outcomes of the RCT will be mental wellbeing, academic stress, comorbid symptoms, and adherence. Analyses will be conducted on an intention-to-treat and per protocol basis.

Discussion: The results of the PROMES-U RCT will provide valuable information on a guided preventive online intervention that could be delivered in the campus context. In addition, results will provide information on the positive impact of the intervention on other relevant factors involved in mental health among university students.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants are all undergraduate students at the 6 participating universities and students followed in the PROMES-U observational study
* Having 18 years of age or more
* Having literacy in Spanish
* Having access to a smartphone (Android or Apple)
* With mild or moderate depression and/or anxiety symptoms screened (i.e., depression (5≤ (PHQ-9) ≤14); and/or anxiety (5≤ GAD-7 ≤14).

Exclusion Criteria:

* Moderately severe or severe depression and/or anxiety (i.e., PHQ-9≥15 and/or GAD-7≥15)
* High suicide risk
* A history of severe psychiatric disorder (e.g., bipolar, psychosis)
* Being on mental health treatment (i.e., medication, psychotherapy or other intervention)

Students with high suicide risk will receive a clinical alert recommending them to visit a specialist and a list of available mental health resources.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change of depressive symptoms | Up to 6 weeks, at 6 months and 12 months after randomization
  The primary outcome will be the change of depressive symptoms at post-intervention (up to 6 weeks), 6 months and 12 months post randomization, considering the minimal clinically relevant change in the scores of Patient Health Questionnaire-9 (PHQ-9) and the Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS).
  The PHQ-9 range from 0 to 27, higher scores mean a worse outcome. The PHQ-ADS range from 0 to 48 with higher scores indicating more severe depression.
Change of anxiety symptoms | Up to 6 weeks and at 6 months and 12 months post randomization
  The primary outcome will be the change of anxiety symptoms at post-intervention (up to 6 weeks), 6 months and 12 months post randomization, considering the minimal clinically relevant change in the scores of Generalized Anxiety Disorder -7 (GAD-7) he Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS).
  The GAD-7 range from 0 to 21, higher scores mean a worse outcome. The PHQ-ADS range from 0 to 48 with higher scores indicating more severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Alonso, Principal Investigator — Hospital de Mar Medical Research Institute (IMIM)
Locations (1):
- Miquel Roca, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ballester L, Gili M, Roca M, Forteza-Rey I, Soto-Sanz V, Vilagut G, Amigo F, Moreno-Kustner B, Mortier P, Piqueras JA, Portillo-Van Diest A, Rebagliato M, Rodriguez-Jimenez T, Alonso J; PROMES-U study group. Effectiveness of a guided mobile app intervention for depression and anxiety in university students (PROMES-U study): protocol of a multicenter randomized controlled trial. BMC Public Health. 2025 Nov 3;25(1):3740. doi: 10.1186/s12889-025-24752-3. PMID 41184908